CLINICAL TRIAL: NCT07344610
Title: Effects of Short-term Intensive Statin Therapy on Lipid Levels in Patients With Ischemic Stroke or Large Artery Atherosclerosis: A Prospective Observational Study
Brief Title: Effects of Short-term Intensive Statin Therapy on Lipid Levels
Status: Recruiting | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Other Study IDs: Y (2025) 527
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: statin — Atorvastatin 40-80mg/day, Rosuvastatin 20mg/day

SUMMARY:
Acute cerebral infarction (ACI), often linked to arterial stenosis, is a major cause of death and disability. Statins are cornerstone therapies for secondary prevention, effectively lowering LDL-C and stabilizing plaques. However, patient response to intensive statin therapy varies significantly. This prospective study aims to analyze the short-term lipid-lowering effects and influencing factors of such therapy in ACI patients with stenosis, to guide personalized treatment and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Diagnosis of ischemic stroke (within 14 days of onset) confirmed by cranial CT/MRI; or imaging-confirmed intracranial/extracranial atherosclerotic stenosis (stenosis rate ≥ 50%);
* Intensive statin therapy (e.g., atorvastatin 40-80 mg/day or rosuvastatin 20 mg/day) initiated within 24 hours of admission, with a planned continuous application for at least one week;
* Signed informed consent form.

Exclusion Criteria:

* Use of statin therapy within 1 week prior to admission;
* Receiving other lipid-lowering treatments;
* Presence of other serious comorbidities (e.g., malignant tumors, end-stage heart failure) with an expected survival of <1 year;
* Pregnant or lactating women;
* Participation in other drug clinical trials within 3 months;
* Other conditions deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with ischemic stroke (within 14 days of onset) confirmed by cranial CT/MRI, or imaging-confirmed intracranial/extracranial atherosclerotic stenosis (stenosis rate ≥ 50%);
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Absolute reduction in Low-Density Lipoprotein Cholesterol | 7±1 days

SECONDARY OUTCOMES:
Absolute and relative reductions in other lipid parameters (Total Cholesterol, Triglyceride, High-Density Lipoprotein Cholesterol, Lipoprotein a) | 7±1 days
Changes in high-sensitivity C-reactive protein | 7±1 days

CONTACTS AND LOCATIONS:
Locations (1):
- Lu Wang, Shenyang, Liaoning, China